CLINICAL TRIAL: NCT06332664
Title: Collaborative Tele-Nutritional Care for Patients With Stage IV Cancer Undergoing Chemotherapy: The Randomised Clinical Trial
Brief Title: Collaborative Tele-Nutritional Care for Patient With Stage IV Cancer
Acronym: T-NICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xingchen Peng (Other)
Responsible Party: Sponsor-Investigator, Xingchen Peng, PhD, Professor, West China Hospital
Organization: West China Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2023-2330
Record Dates: First submitted 2024-03-10; First posted 2024-03-27 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Nutrition
Keywords: cancer cachexia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early Nutrition Intervention (Experimental): For patients meeting the inclusion criteria and randomly assigned to the intervention group, the investigators will assess their nutritional status monthly. During the home-based period between chemotherapy cycles, the investigators will conduct follow-up and provide care using a mobile application (APP). In the event of new nutritional risks emerging in patients, timely recommendations for medical consultation will be made, and nutritional plans will be formulated accordingly.
  Interventions: Combination Product: Early Nutrition Intervention
- standard care (No Intervention): Patients randomly assigned to the standard treatment group will receive standard care for cancer patients and will not be scheduled for interdisciplinary supportive therapy assessment unless requested by the patient, the primary oncologist, or their family.

INTERVENTIONS:
Combination Product: Early Nutrition Intervention — This involves a multidisciplinary team intervention, including oncologists, nutritionists, and nurses. Additionally, the intervention introduces a team-developed mobile application (APP) for the purpose of regular patient follow-ups to identify nutritional risks promptly and facilitate timely interventions. Patients identified as at risk through the app follow-up will be referred to the nutrition clinic for consultation to address nutritional concerns. For advanced-stage cancer patients undergoing monthly chemotherapy hospitalizations, comprehensive assessments encompassing nutrition, psychological aspects, and other facets will be conducted during hospital stays. When deemed necessary, patients will receive dietary guidance and nutritional support.
  Arms: Early Nutrition Intervention

SUMMARY:
In China, the treatment of advanced-stage cancer often follows a pattern where the management of patients is primarily overseen by oncologists who focus on addressing the main clinical symptoms and intervening accordingly.

However, symptoms such as appetite loss, weight loss, and anxiety are often overlooked. It is common for clinical nutritionists to passively enter oncology wards to conduct comprehensive nutritional assessments and develop nutrition plans only when patients exhibit significant malnutrition, upon request from oncologists or patients and their families.

Against this background, the investigators integrated clinical nutritionists into the oncology treatment team and established a proactive nutritional intervention team specifically targeting stage IV cancer patients. This initiative aims to conduct a single-center, open-label, randomized parallel-group prospective study, with the following objectives: 1) to evaluate the impact of this model on the nutritional status, survival, and quality of life of advanced-stage cancer patients, and 2) to further optimize this model for widespread replication in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

1. The patients should be at the range of 18-80 years old, Eastern Cooperative Oncology Group (ECOG) 0-1.
2. The patients should be diagnosed, untreated stage IV cancer patients requiring chemotherapy;
3. The patients should have good cognitive and reading abilities to complete questionnaires;
4. The patients should have ≥3 months expected survival period

Exclusion Criteria:

1. Patients with neurological or psychiatric disorders affecting cognitive function, including central nervous system metastases from tumors;
2. Patients with severe diseases affecting digestion, metabolism, or food intake;
3. Presence of contraindications to chemotherapy;
4. Patients in a cachectic state or refractory cachexia;
5. Patients with PG-SGA score ≥9 points

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2025-08-30 (Actual); Study Completion 2025-08-30 (Actual)

PRIMARY OUTCOMES:
the incidence of cachexia | every month, up to half year
  The definition and classification of cancer cachexia was used by an international consensus [9, 10]: (1) weight loss > 5% over the past 6 months (in the absence of simple starvation), (2) BMI < 20 and any degree of weight loss > 2%, or (3) appendicular skeletal muscle index consistent with sarcopenia and any degree of weight loss > 2%. The assessment of skeletal muscle depletion was used by mid-upper arm muscle area by anthropometry (men < 32 cm2, women < 18 cm2)

SECONDARY OUTCOMES:
body weight | every month, up to half year
  Changes in body weight over 6 months
Nutritional risk and malnutrition status | every month, up to half year
  Nutrition Risk Screening 2002 (NRS2002) ，the minimum value is 0 and maximum value is 7, and higher scores mean a worse outcome.
Nutritional risk and malnutrition status | every month, up to half year
  Patient-Generated Subjective Global Assessment (PG-SGA)，the minimum value is 0 and maximum value is 20, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: XingChen Peng, Ph.D, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan Universit, Chengdu, Sichuan, China